CLINICAL TRIAL: NCT04365686
Title: Reliable and Rapid Smooth Extubation After Ketofol for Induction of General Anesthesia in Laparoscopic Drilling of Polycystic Ovary: A Randomized Controlled Trial.
Brief Title: Smooth Extubation With Ketofol for Induction of General Anesthesia in Laparoscopic Drilling of Polycystic Ovary
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Atef Mohamed Sayed mahmoud, Lecturer, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R83
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Smooth Extubation
Keywords: Ketofol; Propofol; Laparoscopic Drilling of Polycystic Ovary
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group K (Active Comparator): Ketofol group
  Interventions: Drug: Ketofol as induction agent
- Group P (Active Comparator): propofol group
  Interventions: Drug: Propofol as induction agent

INTERVENTIONS:
Drug: Ketofol as induction agent — Patients who received propofol (1mg/kg) plus ketamine (0.5mg/kg) at the induction of general anesthesia
  Arms: Group K
Drug: Propofol as induction agent — Patients who received propofol (2mg/kg) only at the induction of general anesthesia.
  Arms: Group P

SUMMARY:
the effect of ketofol, a combination of propofol and ketamine, on hemodynamics and airway response during induction of general anesthesia has been studied before. Its effect on the smoothness of extubation has not been studied before. In the present study; we aimed to assess the effect of ketofol on the smoothness of extubation as regards, airway response, sedation score during suction and extubation and hemodynamic changes comparing it with propofol for induction of general anesthesia.

DETAILED DESCRIPTION:
After securing intravenous access by a 20g catheter, intravenous premedication (midazolam 2 mg and 4mg ondansetron) was administered to all patients. Standard ASA(american society of anesthesiologists) monitoring (5-lead ECG, noninvasive blood pressure (NIBP), and pulse oximetry) was applied to all the patients for the recording of heart rate (HR), NIBP and oxygen saturation by a multiparameter monitor. Induction of general anesthesia was achieved as follows: in Group K (Ketofol group), fifty three female patients received propofol (1mg/kg) plus ketamine (0.5mg/kg) at the induction of general anesthesia while in Group P (Propofol group), fifty three female patients received propofol (2mg/kg) only at the induction of general anesthesia.

Patients in both groups received fentanyl 2 ug\kg and atracurium 0.5 mg\kg. After tracheal intubation, general anesthesia maintained by isoflurane 1.5 volume % in 2 L\min oxygen-air mixture 50:50 and atracurium 0.1 mg\kg every 30 minutes, if needed. At the end of the surgery, inhalational anesthesia was stopped and reversal of the patients was done by injection of neostigmine 0.05mg\ kg and atropine 0.01mg\kg.

Hemodynamics (HR and mean arterial pressure ''MAP'') was assessed at 5 minutes interval from the time of reversal of muscle relaxant up to 30 minutes after extubation.

The level of sedation during suction and extubation was assessed using observer assessment sedation score and the airway response under direct laryngoscopy to suction was noted by five-point scale. After 5 minute interval, the level of sedation and smoothness of extubation was noted by four-point scale.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Physical status ''ASA PS'' class I and II scheduled for laparoscopic drilling for polycystic ovary under general anesthesia.

Exclusion Criteria:

* from cardiac, hepatic, renal diseases, history of epilepsy
* Patient refusal.
* known drug allergy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — patient with polycystic ovary.
Enrollment: 106 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-12 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
smoothness of extubation | 5 minutes after extubation
  Smoothness of extubation Grade Description
  1. No coughing on endotracheal tube
  2. Coughing on the tube
  3. Vomiting
  4. Laryngospasm

SECONDARY OUTCOMES:
airway response to laryngoscopy and suction | 5 minutes after extubation
  Grading of air way reflexes Grade Description
  1. Excellent(breathing well, no response to laryngoscopy& suctioning)
  2. Good(breathing well, minimal grimacing response to laryngoscope& suctioning)
  3. Satisfactory (breathing well coughing attempt to laryngoscopy& suctioning)
  4. Poor (breathing well, coughing on tube laryngoscopy)
  5. Very poor (breathing well, coughing on tube laryngoscopy)
sedation score | 5 minutes after extubation
  Observer assessment sedation score Observation Score Responds readily to name spoken in normal tone 5 Lethargic response to name spoken in normal tone 4 Responds only after name is called loudly and\or repeatedly 3 Responds only after mild podding or shaking 2 Dose not responds to mild podding or shaking 1
Age | 6 hours before intervention
  In years
weight | 6 hours before intervention
  In kilograms
Height | 6 hours before intervention
  In meters
BMI | 6 hours before intervention
  In kilogram per square meter
mean arterial pressure (MAP) | 5 minutes before extubation
  hemodynamic parameter
mean arterial pressure (MAP) | 1 minute after extubation
  hemodynamic parameter
mean arterial pressure (MAP) | 5 minutes after extubation
  hemodynamic parameter
mean arterial pressure (MAP) | 10 minutes after extubation
  hemodynamic parameter
mean arterial pressure (MAP) | 15 minutes after extubation
  hemodynamic parameter
mean arterial pressure (MAP) | 20 minutes after extubation
  hemodynamic parameter
heart rate (HR) | 5 minutes before extubation
  hemodynamic parameter
heart rate (HR) | 1 minute after extubation
  hemodynamic parameter
heart rate (HR) | 5 minutes after extubation
  hemodynamic parameter
heart rate (HR) | 10 minutes after extubation
  hemodynamic parameter
heart rate (HR) | 15 minutes after extubation
  hemodynamic parameter
heart rate (HR) | 20 minutes after extubation
  hemodynamic parameter

CONTACTS AND LOCATIONS:
Overall Officials: Atef S Khalil, MD, Principal Investigator — Fayoum University Hospitals
Locations (1):
- Fayoum University hospital, Al Fayyum, Madīnat Al Fayyūm, Faiyum Governorate, Egypt, Egypt